CLINICAL TRIAL: NCT02903225
Title: Clinical Value of Heart Rate Variability Indexes to Predict Outcomes After Exercise Training in Chronic Heart Failure
Acronym: REINCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Roberto Ricca-Mallada, Medical Doctor, Magister in Science, Universidad de la Republica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARDIAC REHABILITATION HF
Record Dates: First submitted 2016-09-05; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Heart Failure; Systolic Heart Failure
Keywords: Heart rate variability; Systolic heart failure; Physical exercise; Parasympathetic indexes
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Motor Activity | interventions — Cardiac Rehabilitation; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): usual care and no changes in their previous physical activity
- Cardiac Rehabilitation (Active Comparator): Exercise Training program on a 3-days/week basis during 24 weeks (68-74 sessions). Each session started with a 10-min warm-up walking period followed by 20-min of breathing exercises and free non-resistance movements of limbs. This stage was followed by pedaling during 20-minutes at a circuit resistance training protocol using a stationary cycle-ergometer. Each session ended with a cool down period (5-minutes) including diverse stretching maneuvers of engaged muscle groups. The initial bicycle-ergometer workload (WL) was defined as 50% of the maximum achieved in the previous stress testing
  Interventions: Behavioral: Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — All patients included in this group attended a supervised exercise training program. A cardiologist supervised the hole training sessions. Blood pressure, pulse rate, oxygen saturation, and body weight were measured in each session. The modified Borg scale was used to measure the perceived exercise intensity
  Other Names: Exercise training; Educational approach
  Arms: Cardiac Rehabilitation

SUMMARY:
Controlled exercise training is a valuable therapeutic addition to pharmacological treatment in most patients with chronic heart failure, reducing long-term mortality, preventing cardiac remodeling and improving functional capacity. Despite the mechanism underlying its benefits might be multifactorial, a sustained improvement in autonomic balance is usually attributed as a major effect. Nevertheless, not all eligible subjects show the same response to exercise, probably due to several differences in the subpopulations enrolled. The investigators hypothesize that some Heart Rate Variability indexes could be valid tools to optimize the selection and follow-up of chronic heart failure patients to training

DETAILED DESCRIPTION:
Forty subjects followed in a University Heart Failure Management Program were prospectively included. All patients were evaluated before the randomization and after 24 weeks from enrollment. The investigators performed a detailed anamnesis and complete physical examination, Doppler echocardiography, Stress Testing, 6-minute walk test, heart rate variability analysis, and quality of life test. Patients were randomized either to a training group: performing a supervised training program, or a control group receiving usual care. All patients received an optimal pharmacologic treatment including diuretics, angiotensin converting enzyme inhibitors or angiotensin receptor blockers and beta-adrenergic blocking agents. All patients included in the training group attended a supervised program 3-days/week during 24 weeks (68-74 sessions). Physical aerobic training appears to impart beneficial changes in autonomic control of patients with chronic heart failure through both parasympathetic and sympathetic control of hear rate. These effects produce changes in several Heart Rate Variability indices as HF and rMSSD related with parasympathetic tone.

ELIGIBILITY:
Inclusion Criteria:

* subjects followed in a University Heart Failure Management Program
* maintained sinus rhythm
* New York Heart Association Functional Class (NYHA) I to III and
* LVEF≤40% documented by echocardiogram
* optimal pharmacologic treatment

Exclusion Criteria:

* history of stroke, myocardial infarction or extended anterior myocardial scar
* revascularization procedures or recurrent angina within previous 3 months
* orthopedic impairment
* alcohol or drug abuse;
* implant of pacemaker or cardioverter-defibrillator (AICD);
* frequently ventricular dysrhythmias,
* atrial flutter or fibrillation
* insulin-dependent diabetes mellitus;
* severe chronic obstructive pulmonary disease or renal dysfunction
* comorbid non-cardiac disease limiting short term survival
* previous enrollment in an ET program
* subjects at great propensity for noncompliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clinical Events | 6 month
  Change in New York Heart Association Functional Class; Number of hospitalizations 6 months before and after the date of enrollment; temporary or permanent withdrawal from the study protocol (due to persistent atrial or ventricular arrhythmias; worsening of congestive heart failure symptoms; myocardial infarction; unstable angina; need of cardiac interventions: pacemaker, implantable cardioverter defibrillator, coronary revascularization or cardiac transplantation; stroke or transient ischemic attack; severe peripheral intermittent claudication or death observed during training or follow-up sessions
Mean heart rate | 6 month
  the mean value of the12-min Electrocardiogram-recordings was considered the resting heart rate (beats per minute)
6 minute walk test | 6 month
  walking along a 20-meter long corridor at their own pace, with the aim of covering as much ground as possible in 6 minutes. The distance walked was expressed in meter
left ventricular ejection fraction | one year
  The area-length method was measured to obtain biplane left ventricle volumes. Left Ventricle ejection fraction was derived from the standard equation (%)
quality of life | 6 month
  All the subjects completed the Short-Form 36 Health Survey (SF-36), available in its Spanish version, for measuring physical and mental quality of life
Stress Test | 6 month
  symptom limited exercise testing, measured in metabolic unit (MET)
square root of the mean squared successive differences of R-R intervals (rMSSD) | 6 month
  short-term continuous electrocardiographic recordings were performed for heart rate variability analysis. In the time domain, the square root of the mean squared successive differences of R-R intervals (rMSSD) were calculated. Units: ms
Heart rate power high-frequency (HF) | 6 month
  The high-frequency (HF), from 0.15 to 0.40 Hz of the power spectral analysis were calculated. Units: ms2/Hz

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Ricca-Mallada, MD MSc, Principal Investigator — Hospital de Clinicas

IPD SHARING:
Plan to Share IPD: No